CLINICAL TRIAL: NCT02611453
Title: CO2 Cholangiography as an Alternative to Iodinated Contrast in Endoscopic Retrograde Cholangiopancreatography
Brief Title: Cholangiography Using Carbon Dioxide Versus Iodinated Contrast in ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Andrew Y Wang, MD, Associate Professor of Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18285
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Choledocholithiasis; Bile Duct Diseases; Bile Duct Carcinoma
Keywords: choledocholithiasis; ERCP; cholangiography; biliary stricture; bile ducts; carbon dioxide
MeSH Terms: conditions — Choledocholithiasis; Bile Duct Diseases; Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): All patients will undergo endoscopic retrograde cholangiopancreatography (ERCP) that is indicated for suspected or confirmed choledocholithiasis or biliary strictures. "Air" contrast cholangiography using carbon dioxide gas will be performed with standard fluoroscopy and digital subtraction fluoroscopic image capture followed by routine cholangiography using iodinated contrast and standard fluoroscopy. Carbon dioxide (CO2) is routinely used in ERCP procedures and would flow into the biliary tree of patients at the time of ERCP, irrespective of this study's interventions. Digital subtraction image capture is a commercially available setting on certain fluoroscopy units that optimizes resolution with air or CO2 used as a contrast medium.
  Interventions: Other: "Air" contrast cholangiography using carbon dioxide gas

INTERVENTIONS:
Other: "Air" contrast cholangiography using carbon dioxide gas — Carbon dioxide (CO2) will be injected into the biliary tree (which is already exposed to CO2 during routine ERCP) and images will be obtained by using fluoroscopy and digital subtraction imaging (a specific setting on certain fluoroscopy tables).

SUMMARY:
Carbon dioxide (CO2) gas is widely used for luminal insufflation during endoscopic retrograde cholangiopancreatography (ERCP) of the biliary tract. While frequently observed during routine ERCP, there are few data on the topic of "air" or "CO2" cholangiography. Our primary aim is to compare radiographic cholangiograms in patients with biliary tract disease (from stones or strictures) during ERCP obtained by using carbon dioxide as the contrast medium vs. conventional iodinated contrast.

DETAILED DESCRIPTION:
It has been recommended that endoscopic retrograde cholangiopancreatography (ERCP) be performed using carbon dioxide (CO2) instead of room air as the infused "air" or gas for luminal insufflation for reasons of improved patient comfort and in case of procedural adverse events (as CO2 is more quickly absorbed by the body and as it can be exhaled via the lungs). Air cholangiograms are often incidentally visible on fluoroscopy (radiographically) during ERCP prior to injection of iodinated contrast into the biliary tree. Despite the information from an air cholangiogram being readily available in many instances, biliary endoscopists and radiologists who read the fluoroscopic images taken during ERCP do not usually comment or interpret the "air" or "CO2" cholangiograms. Consequently, very little data is available on the topic of "air" or "CO2" cholangiography. As a contrast medium for cholangiography, CO2 might be safer than iodinated contrast, which is the standard contrast medium used during ERCP, as iodinated contrast cannot be easily absorbed by the body and as it can be trapped proximal to obstructing biliary stones or strictures and lead to biliary tract infection.

This is a prospective cohort study that will enroll patients undergoing ERCP for suspected choledocholithiasis and/or biliary stricture(s). If they did not participate in this study, these patients would still require an ERCP with CO2 used as the endoscopically insufflated "air" medium. Enrolled patients will undergo an initial cholangiogram with CO2 (injected into the bile ducts) utilizing both conventional fluoroscopy and digital subtraction fluoroscopic imaging, followed by conventional cholangiography using iodinated contrast (injected into the bile ducts). Digital subtraction fluoroscopic imaging is a commercially available setting on certain fluoroscopy units that optimizes resolution with air or CO2 used as a contrast medium. Findings on CO2 cholangiography will be compared to those obtained from pre-procedural abdominal imaging along with the cholangiogram done using iodinated contrast at the time of the ERCP procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients with choledocholithiasis, benign biliary strictures, malignant biliary strictures
* Biliary pathology suggested or confirmed by imaging with abdominal ultrasonography, CT scan, MRI/MRCP scan, or endoscopic ultrasonography (EUS)

Exclusion Criteria:

* Pregnancy (self reported)
* Presence of cholangitis before ERCP
* Prior history of surgery on the stomach or duodenum that precludes conventional ERCP or prior biliary tree surgery (not including cholecystectomy)
* Failure to selectively cannulate the bile duct
* Life expectancy less than 30 days
* Prisoners
* Patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Technical success of CO2 cholangiography vs. iodinated contrast | Intraprocedural/immediate (during ERCP)
  For choledocholithiasis: correct identification of the number and location of stones. For biliary strictures: correct identification of number and location of strictures.

SECONDARY OUTCOMES:
Technical success of digital subtraction fluoroscopy vs. traditional fluoroscopy (while using CO2 as the contrast medium) | Intraprocedural/immediate (during ERCP)
  For choledocholithiasis: correct identification of the number and location of stones. For biliary strictures: correct identification of number and location of strictures.
Radiation usage/exposure of CO2 cholangiography using conventional fluoroscopy or digital subtraction fluoroscopy vs. iodinated contrast | Intraprocedural/immediate (during ERCP)
  Fluoroscopy/radiation usage/exposure will be measured for each imaging modality and then compared

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Y. Wang, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang R, Zhao L, Liu Z, Wang B, Hui N, Wang X, Huang R, Luo H, Fan D, Pan Y, Guo X. Effect of CO2 cholangiography on post-ERCP cholangitis in patients with unresectable malignant hilar obstruction - a prospective, randomized controlled study. Scand J Gastroenterol. 2013 Jun;48(6):758-63. doi: 10.3109/00365521.2013.779745. Epub 2013 Apr 29. PMID 23621432
- [Background] Pisello F, Geraci G, Modica G, Sciume C. Cholangitis prevention in endoscopic Klatskin tumor palliation: air cholangiography technique. Langenbecks Arch Surg. 2009 Nov;394(6):1109-14. doi: 10.1007/s00423-009-0548-y. Epub 2009 Aug 26. PMID 19707784